CLINICAL TRIAL: NCT05497024
Title: Older Men's Decision Making About Active Surveillance for Prostate Cancer - Aim 3: Decision Aid Cognitive and Usability Testing
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0375; NCI-2022-06569 (Other: Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surveys: Participants may answer questions that are sensitive in nature.
  Interventions: Behavioral: Surveys
- Interviews: The interview may occur over phone, web conferencing, or in-person.
  Interventions: Behavioral: Interviews

INTERVENTIONS:
Behavioral: Interviews — Participants will discuss background, such as race, education, and living situation.
  Participants will discuss Prostate cancer Participants will discuss feedback on the educational material
  Groups: Interviews
Behavioral: Surveys — Participants may answer questions that are sensitive in nature.
  Groups: Surveys

SUMMARY:
This protocol describes development and user testing of an educational shared decision making intervention to help men with prostate cancer who are on active surveillance make decisions with their health care providers about if and when to de-escalate surveillance testing. The project is important because for many patients their cancer does not progress to the point of needed curative treatment or their health status changes such that they are no longer good candidates for treatment. For these men, de-escalating ongoing surveillance (e.g., fewer biopsies or imaging studies) is a reasonable option.

DETAILED DESCRIPTION:
Objectives:

The overall goal of this protocol is to develop and refine an educational tool for use by patients and health-care providers to help men with localized prostate cancer make informed decisions about discontinuation of active surveillance.

* Conduct cognitive and initial usability and acceptability testing of a prototype decision aid with patients
* Conduct cognitive and initial usability and acceptability testing of a prototype decision aid with care partners/caregivers
* Conduct expert reviews of a prototype decision aid with clinicians

ELIGIBILITY:
Patients

Inclusion Criteria:

1. Males aged 65 or older
2. Diagnosis of localized prostate cancer
3. On active surveillance for 12 or more months
4. Fluent in English

Exclusion Criteria:

1. Receiving treatment for another cancer (primary or recurrence)

Caregivers

Inclusion Criteria:

1. Aged 18 or older
2. Fluent in English
3. Involved with the care of an eligible patient (i.e. partner, close friend, family member, companion)

   Exclusion Criteria:
4. None

Clinicians

Inclusion Criteria:

1. Aged 18 or older
2. Fluent in English
3. Provides clinical care for patients with prostate cancer (e.g. medical oncologists, urologists, radiation oncologists, nurse practitioners, physician assistants)

Exclusion Criteria:

1. None

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Male
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
The Ottawa Acceptability Scale | through study completion and average of 1 year
  The Ottawa Acceptability scale includes 10 items to assess participant's rating of the educational material ease of use, clarity of information, length, level of detail provided, ability to hold one's interest, and satisfaction with how the materials prepared them for discussing the decision with their clinician
  Score Scale (Strongly agree, Agree, Neither agree nor disagree, Disagree Strongly disagree) and (Not at all, A little, Somewhat, Quite a bit, A great deal)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lowenstein, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org